CLINICAL TRIAL: NCT04032990
Title: Transcutaneous Spinal Stimulation Promoting Recovery of Hand and Arm Function After Pediatric-onset Spinal Cord Injury
Brief Title: Transcutaneous Spinal Stimulation: Safety and Feasibility for Upper Limb Function in Children With Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: The Jewish Heritage Foundation for Excellence (Unknown)
Responsible Party: Principal Investigator, Andrea L. Behrman, PhD, PT, Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 19.0810
Record Dates: First submitted 2019-07-16; First posted 2019-07-25 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Spinal Cord Injuries
Keywords: pediatric-onset; transcutaneous spinal stimulation; upper extremity function
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Transcutaneous spinal stimulation - Acute and Training (Experimental): Safety and feasibility outcome measures are collected during application of transcutaneous spinal stimulation while upper extremity function is assessed at 3 time points (acute) and/or in combination with activity-based upper extremity training (40 sessions, 1.5 hours/day, 5 days/week); stimulation will be applied intermittently for no more than 10 minutes at a time. Upper extremity training is based on usual care activities to challenge use of the hands and arms, e.g. reaching, grasping, manipulating objects.
  Interventions: Device: Biostim-5 transcutaneous spinal stimulator

INTERVENTIONS:
Device: Biostim-5 transcutaneous spinal stimulator — Safety and feasibility will be monitored during transcutaneous spinal stimulation in children with spinal cord injury

SUMMARY:
Children who suffer a spinal cord injury in the neck region have difficulty using their hands due to paralysis and/or weakness of their arms and hand muscles. The purpose of this project is to test the safety, comfort, and practicality of a new therapy that stimulates the spinal cord to facilitate activation of arm and hand muscles while practicing grasping, pinching, and reaching movements. The long-term goal is to provide better therapies that will improve the ability of children with SCI to more successfully play and accomplish everyday tasks using their arms and hands, similar to before their injury.

DETAILED DESCRIPTION:
Adults with cervical spinal cord injury (SCI) rank gaining arm and hand function as the highest priority for improving their quality of life. Children with SCI, similarly experience paralysis of hand and arm muscles that limits their engagement in play and exploration typical for child development . Furthermore, pediatric-onset SCI disrupts the acquisition of motor skills involved in activities of daily living such as feeding, dressing and grooming increasing the child's dependence on a parent/caregiver. Current interventions teach persons with SCI to use a brace or splint to compensate for paralysis or weakness of hand muscles. Others are invasive requiring nerve or tendon transplantation and/or electrode implantation for functional electrical stimulation. Transcutaneous electrical spinal cord stimulation (TcStim) is a non-invasive painless technique that augments the intrinsic capacity of the spinal cord below the level of injury to generate patterned motor output. In adults with chronic SCI, TcStim acutely (immediately) augments trunk control and improves upper extremity function when combined with task-specific training. In children with cerebral palsy, TcStim in combination with locomotor training improves walking ability. Thus, the long-term objectives are 1) to investigate the therapeutic potential of TcStim for improving arm/hand function and 2) provide high quality scientific evidence to guide the clinical use of neurotherapeutic interventions promoting recovery in children with SCI. As children with SCI represent a vulnerable population, we first must establish the safety and feasibility of any potential novel therapeutic approach. Therefore, the specific aims of this proposal are to 1) determine proof-of-principle, safety and feasibility of TcStim for acute increase of hand/arm function in children with SCI and 2) determine the safety and feasibility of TcStim in combination with activity-based upper extremity training (AB-UET) across 40 sessions in children with SCI. For this pilot study 8-10 participants, ages 5-18 years with chronic, acquired SCI who have completed ≥ 40 sessions of activity-based upper extremity training (AB-UET) with neuromuscular stimulation will be recruited. For Aim 1, TcStim parameters will be optimized for arm/hand function. Arm/hand function will be assessed using the three tasks: overhead reach, forward reach and grasp and in-hand manipulation for no-TcStim and TcStim conditions measuring kinematics, electromyography of arm and hand muscles. For Aim 2 (safety and feasibility), two participants will undergo 40 sessions of AB-UET in combination with TcStim. To assess long-term safety and feasibility, participant compliance and any difficulties (i.e. risks, discomfort) will be documented and risk-likelihood/risk-benefit established. The long-term goal is to provide better therapies that will improve the ability of children with SCI to use their arms and hands with more success to grasp, reach and use their hands for everyday play and daily tasks.

ELIGIBILITY:
Inclusion Criteria:

* history of chronic, acquired SCI, (>1 year since injury);
* SCI involves cervical and/or high thoracic (T1) levels
* moderate to severe upper extremity deficit as assessed by the Pediatric Neuromuscular Recovery Upper Extremity Scale (scores less than 4A out of a 12 point range from 1A-4C on upper extremity tasks, e.g. including inability to fully reach overhead, grasp, or pinch without compensation)
* discharged from in-patient rehabilitation

Exclusion Criteria:

* botox use within past 3 months;
* current baclofen use
* unhealed upper extremity fracture
* any other medical complication limiting participation in the assessments and/or activity- based upper extremity training;
* congenital SCI
* total ventilator dependence

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-11-14 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of skin irritation | within 2 months for Aim 1, within 3 months for Aim 2
  Skin color, particularly change in skin color to pink indicating irritation in the location of the stimulating electrode placement will be assessed prior to stimulation experiments and immediately after; incidence of pink- or redness or irritation and time (minutes-days) to dissipation will be recorded.
Faces Pain Scale-Revised (scale 0-10) | within 2 months for Aim 1, within 3 months for Aim 2
  Faces Pain Scale - Revised is a self-report measure of pain intensity developed for children (C.L. Hicks et al. Pain 93 (2001). It will be used to score the sensation of pain on 0 (min - no pain)-to-10 (max - worst pain ever) metric. The scale depicts 6 facial expressions: first - face with a neutral expression corresponds to pain score of 0, next facial expression is scored as 2, etc. The faces scale will be presented to the participant (ages 3-8) prior to the experiment for baseline measurement, during stimulation and following the experiment.
Visual Analog Scale (0-10) | within 2 months for Aim 1, within 3 months for Aim 2
  To assess pain in the participants ages 8 and above, Visual Analog Scale (self-reported measure) will be presented with 0 corresponding to no pain and 10 corresponding to the "worst pain ever"; the scale will be presented at baseline measurement, during stimulation and following the experiment.
Blood pressure | within 2 months for Aim 1, within 3 months for Aim 2
  continuous beat-by-beat blood pressure (mmHg) recordings will be made using Finapres finger cuff system for 5 minutes prior to and 5 minutes immediately following stimulation while the child is sitting; Brachial arm blood pressure will be periodically measured during stimulation (mmHg).
  systolic and diastolic blood pressure values will be compared with the established norms for typically developing children (age and height matched);
Number of requests to stop the stimulation | within 2 months for Aim 1, within 3 months for Aim 2
  Number of participants requesting (or number of request per participant within experimental sessions) to stop stimulation due to pain, fatigue or any other reason (documented)
Angular excursions of upper extremity and hand | within 2 months for Aim 1, within 3 months for Aim 2
  degrees of flexion/extension, adduction/abduction in elbow, shoulder, wrist, fingers
Hand Grip strength | within 2 months for Aim 1, within 3 months for Aim 2
  A hand grip strength dynamometer will be used to assess strength (Newton)

SECONDARY OUTCOMES:
Heart Rate | within 2 months for Aim 1, within 3 months for Aim 2
  heart rate (beats per minute) will be continuously monitored and recorded using 3-lead electrocardiogram.
Compliance rate | within 2 months for Aim 1, within 3 months for Aim 2
  Compliance - number of sessions missed and reason, willingness to continue participation.
Angular excursions of trunk during trunk control assessments | within 2 months for Aim 1, within 3 months for Aim 2
  trunk kinematics (degrees of flexion/extension) in cervical, thoracic and lumbar regions;

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L Behrman, PT, PhD, Principal Investigator — University of Louisville
Locations (1):
- Department of Neurosurgery, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singh G, Keller A, Lucas K, Borders C, Stout D, King M, Parikh P, Stepp N, Ugiliweneza B, D'Amico JM, Gerasimenko Y, Behrman AL. Safety and Feasibility of Cervical and Thoracic Transcutaneous Spinal Cord Stimulation to Improve Hand Motor Function in Children With Chronic Spinal Cord Injury. Neuromodulation. 2024 Jun;27(4):661-671. doi: 10.1016/j.neurom.2023.04.475. Epub 2023 Jun 1. PMID 37269282